CLINICAL TRIAL: NCT07062198
Title: A Phase 3, Randomised, Double-blinded, Placebo-controlled Study to Evaluate the Efficacy, Tolerability, and Safety of Combined Metabolic Activator Supplementation in Subjects Diagnosed With Alzheimer's Disease
Brief Title: Combined Metabolic Activator Supplementation in Subjects Diagnosed With Alzheimer's Disease
Acronym: COGNIS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ScandiBio Therapeutics AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SB-AD-002
Record Dates: First submitted 2025-06-11; First posted 2025-07-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Collagen; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental)
  Interventions: Drug: Combined metabolic activators
- Placebo Arm (Placebo Comparator)
  Interventions: Other: Collagen and maltodextrin

INTERVENTIONS:
Drug: Combined metabolic activators — A total of 20g of CMA2 with strawberry aroma and colouring agent will be given. The IMP will be provided as a soluble powder packed as individual dosages in identical sachets. The powder should be dissolved in 200 ml preferably cold water before use. The powder can also be used on yoghurt or other food. The subjects will take two daily oral doses of the IMP, one dose just after breakfast and one dose just after dinner. Subjects who cannot tolerate (e.g., diarrhoea) taking full dose will be withdrawn from the study.
  Arms: Treatment Arm
Other: Collagen and maltodextrin — As placebo, a total of 20g of compound primarily containing collagen and maltodextrin will be administered. Placebo contains strawberry aroma flavouring and colouring agent.
  Arms: Placebo Arm

SUMMARY:
This randomised, double-blinded, placebo-controlled study aims to establish metabolic improvements in subjects diagnosed with Alzheimer's Disease (AD) by treatment with CMA2 including N-acetyl-L-cysteine (NAC), L-carnitine-L-tartrate (LCAT), nicotinamide (niacinamide), and L-serine.

Participants will take the drug CMA2 or a placebo twice a day for 26 weeks. They will visit the clinic 4 times for checkups and tests.

DETAILED DESCRIPTION:
This will be a randomised, double-blinded, placebo-controlled, multi-centre Phase 3 study with the aim to establish metabolic improvements in subjects diagnosed with AD by dietary supplementation with CMA2, including NAC, LCAT, niacinamide, and L-serine. The study will be performed at approximately 9 clinical sites in Turkey and aims to include a total of 676 evaluable subjects (up to 845 randomised).

The study comprises four clinical visits. Consenting subjects will be screened for eligibility (Visit 1; screening) according to study-specific eligibility criteria within 28 days prior to randomisation and start of IMP administration. Eligible subjects will be randomised on Day 1 (Visit 2) to 26 weeks of b.i.d. oral administration of either CMA2 or placebo (1:1). The first dose will be administered at the study clinic. The subjects will be observed for 2 hours post dose for the development of any allergic reactions or intolerance after taking the first dose. Subjects who cannot tolerate the study agents will be withdrawn from the study.

Visits at the study site will be performed at Week 13 (Visit 5) and Week 26 (Visit 8; end of treatment). Monthly telephone contacts will be scheduled with the patients. At the telephone visits IMP compliance, Concomitant medication and adverse event will be addressed.

The following clinical scales will be used to assess the effect of CMA2 on cognition and daily life activity: MMSE, ADAS-Cog, and ADCS-ADL. Blood samples will be collected for advanced plasma metabolomics, proteomics, and lipidomics analysis. Whole genome sequencing will not be performed.

Optional blood samples will be collected for p- tau217, Nfl, GFAP, and S-Urate analysis. Optional Saliva and faeces sampling for oral and gut microbiome will be collected. CSF samples will be optional collected for determination of Abeta42, total-Tau, p-Tau181 levels and Neurofilament light chain concentrations, and for advanced CSF metabolomics, proteomics, and lipidomics analysis. These samples will be decided by each investigator and will be analysed as exploratory endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women of non-childbearing potential ≥ 50 years of age.
2. Diagnosed with AD and at the Screening visit having the scores of ADAS-Cog ≥ 12 and GDS≥ 4.
3. Stable AD treatments and clinical course for at least 1 month.
4. Females of childbearing potential must have documented tubal ligation or hysterectomy; or be post-menopausal (defined as 12 months of amenorrhoea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) 25-140 IE/L and oestradiol <200 pmol/Lis confirmatory]).
5. Able to give written informed consent for participation in the study by the patient and/or legal representatives.

Exclusion Criteria:

1. History of stroke.
2. History of brain trauma < 14 days.
3. Uncontrolled diagnosed depression.
4. Uncontrolled (HbA1C > 8) type 1 or type 2 diabetes.
5. Severe swallowing problems.
6. PEG-feeding.
7. Chronic diarrhoea.
8. Chronic kidney disease with S-Creatinin > 1,30 mg/dl.
9. Active bronchial asthma at the time of screening.
10. History of phenylketonuria (contraindicated for NAC).
11. Known allergy for substances used in the study.
12. Known malignancies.
13. Use of dietary supplements such as vitamins, omega-3 products, or plant stanol/sterol products later than one (1) week prior to inclusion.
14. Use of anti-microbial agents later than one (1) week prior to inclusion.
15. Drug and/or alcohol abuse.
16. Subjects considered as inappropriate for this study for any reason (noncompliance etc.) per investigator assessment.
17. Administration of another new chemical entity (defined as a compound that has not been approved for marketing) or has participated in any other clinical study that included drug treatment with the last administration within 3 months prior to administration of IMP in this study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 845 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-Cog) score from baseline to end-of-treatment | Visit 1, Visit 5 (13 weeks), Visit 8 (26 weeks)
  The test administrator adds up points for the errors in each task for a total score ranging from 0 to 70. The greater the dysfunction, the greater the score. A score of 70 represents the most severe impairment and 0 represents the least impairment

SECONDARY OUTCOMES:
Change in Mini Mental State Examination (MMSE) score from baseline to end-of-treatment | Visit 1, Visit 5 (13 weeks), Visit 8 (26 weeks)
  MMSE is administered serially to assess the effect of time on the progression of dementia. The MMSE contains seven domains (including orientation, attention, recall) each with an assigned point value totaling 30. Severe cognitive impairment is indicated by a score of (≤9 points) moderate (10- 20 points) and mild (21-24 points). A score of 25 and over indicates normal cognition.
Change in Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) score from baseline to end-of-treatment | Visit 1, Visit 5 (13 weeks), Visit 8 (26 weeks)
  The 23 ADL items (Activities of Daily Living; 6 basic and 17 instrumental) assess the competence of patients with Alzheimer's Disease in activities of daily living. All responses should relate to the 4 weeks prior to the time of rating. The total score is 0-78, with low scores indicating more severe impairment.
To evaluate compliance daily two doses treatment in patients | Visit 5 (13 weeks), Visit 8 (26 weeks)
  The subject will be instructed to bring all unused IMP and empty containers to the clinic visits on Week 13 and Week 26.
Change in body weight from baseline through-out the study | Visit 1, Visit 5 (13 weeks), Visit 8 (26 weeks)
  Body weight will be measured at Visit 1, Visit 5 and Visit 8 to evaluate the safety of metabolic cofactor supplementation.
Change in body height from baseline through-out the study | Visit 1, Visit 5 (13 weeks), Visit 8 (26 weeks)
  Body height will be measured at Visit 1, Visit 5 and Visit 8 to evaluate the safety of metabolic cofactor supplementation.
Change in BMI from baseline through-out the study | Visit 1, Visit 5 (13 weeks), Visit 8 (26 weeks)
  BMI will be assessed at Visit 1, Visit 5 and Visit 8 to evaluate the safety of metabolic cofactor supplementation.
Change in waist and hip circumference from baseline | Visit 1, Visit 5 (13 weeks), Visit 8 (26 weeks)
  Waist and hip circumference will be measured aat Visit 1, Visit 5 and Visit 8 to evaluate the safety of metabolic cofactor supplementation.
Change in blood pressure from baseline | Visit 1, Visit 5 (13 weeks), Visit 8 (26 weeks)
  Systolic and Diastolic Blood Pressure (mmHg) will be measured at Visit 1, Visit 5 and Visit 8 to evaluate the safety of metabolic cofactor supplementation.
Change in heart rate from baseline | Visit 1, Visit 5 (13 weeks), Visit 8 (26 weeks)
  Change in heart rate will be measured at Visit 1, Visit 5 and Visit 8 to evaluate the safety of metabolic cofactor supplementation
Change in red blood cell count from baseline | Visit 1, Visit 5 (13 weeks), Visit 8 (26 weeks)
  Red Blood Cell count test will be performed to measure possible toxic effects of metabolic cofactor supplementation on the hematological system.
Change in platelet count from baseline | Visit 1, Visit 5 (13 weeks), Visit 8 (26 weeks)
  Platelet count test will be performed to measure possible toxic effects of metabolic cofactor supplementation on the hematological system.
Change in hemoglobin concentration from baseline | Visit 1, Visit 5 (13 weeks), Visit 8 (26 weeks)
  Hemoglobin concentrations will be assessed to measure possible toxic effects of the metabolic cofactor supplementation on hematological system.
Change in white blood cell count from baseline | Visit 1, Visit 5 (13 weeks), Visit 8 (26 weeks)
  White blood cell count test will be performed to measure possible toxic effects of the metabolic cofactor supplementation on hematological system.
Changes in kidney function tests from baseline | Visit 1, Visit 5 (13 weeks), Visit 8 (26 weeks)
  Kidney function tests (creatinine, urea, urate) will be performed to measure possible toxic effects of the metabolic cofactor supplementation on kidney function.
Changes in kidney function tests from baseline | Visit 1, Visit 5 (13 weeks), Visit 8 (26 weeks)
  Kidney function tests (sodium, potassium) will be performed to measure possible toxic effects of the metabolic cofactor supplementation on kidney function.
Changes in liver function tests [Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Gamma-glutamyl transferase (GGT), Alkaline phosphatase (ALP)] from baseline | Visit 1, Visit 5 (13 weeks), Visit 8 (26 weeks)
  Liver function tests (ALT, AST, GGT, ALP) will be performed to measure possible toxic effects of the metabolic cofactor supplementation on liver function.
Changes in liver function tests (Total Bilirubin, and Albumin) from baseline | Visit 1, Visit 5 (13 weeks), Visit 8 (26 weeks)
  Liver function tests (Total Bilirubin, Albumin) will be performed to measure possible toxic effects of the metabolic cofactor supplementation on liver function.
Changes in creatinine kinase (CK) level from baseline | Visit 1, Visit 5 (13 weeks), Visit 8 (26 weeks)
  Creatinine kinase (CK) level will be evaluated to measure possible toxic effects of the metabolic cofactor supplementation.
Changes in blood lipid levels (total cholesterol (TC), triglyceride (TG), low density lipoprotein (LDL-C), high density lipoprotein (HDL-C)) from baseline | Visit 1, Visit 5 (13 weeks), Visit 8 (26 weeks)
  Blood lipid levels (total cholesterol (TC), triglyceride (TG), low density lipoprotein (LDL-C), high density lipoprotein (HDL-C)) will be evaluated to measure possible toxic effects of the metabolic cofactor supplementation.
Changes in blood glucose levels from baseline | Visit 1, Visit 5 (13 weeks), Visit 8 (26 weeks)
  Blood glucose levels will be evaluated to measure possible toxic effects of the metabolic cofactor supplementation.
Change in blood insulin level from baseline | Visit 1, Visit 5 (13 weeks), Visit 8 (26 weeks)
  Blood insulin level will be evaluated to measure possible toxic effects of the metabolic cofactor supplementation.
Change in thyroid-stimulating hormone (TSH) level from baseline | Visit 1, Visit 5 (13 weeks), Visit 8 (26 weeks)
  Thyroid-stimulating hormone (TSH) level will be evaluated to measure possible toxic effects of the metabolic cofactor supplementation.
Monitoring Adverse Events | 26 weeks
  This process aiming to monitoring of adverse events of metabolic cofactor supplementation. Adverse events, serious adverse events, serious adverse reactions, suspected unexpected serious adverse reactions will be monitored continuously and all events that occur at any time during the study will be reported in Case Report Forms. Any symptoms of intestinal discomfort or other side effects will be carefully recorded and all study subjects will be informed to contact (by phone or text message) the investigators immediately if they experience any symptoms of discomfort or any side effects during the intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Sevki SAHIN, Prof. Dr., Principal Investigator — Sancaktepe Şehit Prof. Dr. İlhan Varank Training and Research Hospital, University of Health Sciences Istanbul 34766, Turkiye
Locations (8):
- Turkey (Türkiye) (8):
  - Department of Neurology and Neuroscience, Faculty of Medicine, Alaaddin Keykubat University, Alanya
  - Ataturk University, Faculty of Medicine, Department of Neurology, Erzurum, Turkey; Movement Disorders and Neuromodulation Center, Ataturk University, Erzurum
  - Behavioural Neurology and Movement Disorders Unit, Department of Neurology, Istanbul Faculty of Medicine, Istanbul University, Istanbul
  - Haydarpaşa Numune Training and Research Hospital, University of Health Sciences Istanbul, Istanbul
  - Sancaktepe Şehit Prof. Dr. İlhan Varank Training and Research Hospital, University of Health Sciences Istanbul, Istanbul
  - SB Haseki Training and Research Hospital, Istanbul, University of Health Sciences Istanbul, Istanbul
  - Sultan Abdülhamid Han Training and Research Hospital, University of Health Sciences Istanbul, Istanbul
  - Umraniye Training and Research Hospital, University of Health Sciences Istanbul, Istanbul

IPD SHARING:
Plan to Share IPD: No